CLINICAL TRIAL: NCT01897285
Title: A Single Centre, Randomised, Comparative, Blinded Wear Test of Two Adhesives on the AQUACEL® Foam Adhesive Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: CW-0209-13-U368
Record Dates: First submitted 2013-05-10; First posted 2013-07-11 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Safety and Performance of Dressing Adhesive on Healthy Volunteers
Keywords: Performance and safety of the AQUACEL® foam adhesive dressing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- All study participants: AQUACEL® foam adhesive dressings (Experimental): Original adhesive + test adhesive
  Interventions: Device: AQUACEL® foam adhesive dressing

INTERVENTIONS:
Device: AQUACEL® foam adhesive dressing

SUMMARY:
AQUACEL® foam adhesive dressing is a sterile Hydrofiber® foam wound dressing consisting of a waterproof outer polyurethane film, and a multi-layered absorbent pad, having a silicone adhesive border. The multi-layered absorbent pad contains a layer of polyurethane foam and a non-woven wound contact layer of Hydrofiber® (NaCMC). This dressing product was launched in 2012. A new source of silicone adhesive is now under assessment for this product. This Healthy Volunteer Wear test will form part of the Design Validation for this change in supplier and is required to confirm that the new Silicone Adhesive trilaminate supplier can coat the silicone adhesive to provide comparable adhesive dressing performance in terms of wear time, ease of use and with a similar safety profile in relation to the skin.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Be a healthy volunteer and be over 18 years of age
* Be willing to attend two scheduled visits for application and removal of the device and adverse event review
* Have healthy unbroken skin

Exclusion Criteria:

* Subjects with a history of sensitivity to any one of the components of the device being studied
* Female subjects who are currently pregnant or lactating
* Subjects who are not willing and able to attend the 'clinic' for the required assessments
* Subjects with excessive hair on their backs
* Subjects who have any other medical condition which, according to the investigator justifies exclusion from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Lawrence, RGN, Principal Investigator — Wirral University Teaching Hospital NHS Trust
Locations (1):
- Global Development Centre, Deeside Industrial Park, Deeside, Flintshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Original adhesive and Test adhesive on right and left upper arm and right and left lower back.
  AQUACEL® foam adhesive dressing Original Adhesive: Arm, Test Adhesive: Arm, Original Adhesive: Back, Test Adhesive: Back
Period: Overall Study
Arm/Group | All Study Participants
Started | 20 (All 20 participants received original AND test adhesive dressings on upper arms and lower back.)
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Ten male (50%) and ten female (50%) healthy volunteers were enrolled into the study with a mean age of 37.1 years.
Groups:
- All Participants: AQUACEL® Foam Adhesive Dressings: Original adhesive + test adhesive
  AQUACEL® foam adhesive dressings
Arm/Group | All Participants: AQUACEL® Foam Adhesive Dressings
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Product Performance (Adhesion, Conformability, Ease of Application/Removal, Adhesive Residue, Comfort During Removal, Condition of the Skin)
Description: * Adhesion at 7 days measured by:
    1 = Excellent 2 = Good 3 = Average 4 = Poor 5 = Very Poor
  * Conformability
    1 = Excellent 2 = Good 3 = Average 4 = Poor 5 = Very Poor
  * Dressing Integrity
    1 = Excellent 2 = Good 3 = Average 4 = Poor 5 = Very Poor
  * Ease of Application
    1 = Excellent 2 = Good 3 = Average 4 = Poor 5 = Very Poor
  * Ease of Removal,
    1 = Very easy 2 = Easy 3 = Difficult 4 = Very difficult
  * Adhesive Residue 0 = None 1 = Minimal 2 = Moderate 3 = Considerable
  * Comfort during removal
    1 = Excellent 2 = Good 3 = Average 4 = Poor 5 = Very Poor
  * Condition of the skin This will be evaluated by the Skin Irritation Scale (Doubtful reaction/weak positive reaction/ strong positive reaction/ extreme positive reaction/irritant reaction/ negative reaction)
Time Frame: 7 days
Population: 20/20 subjects completed maximum study participation of 7 days. Two subjects dressings detached very early on so returned for their final evaluation on the second day. The final subject status was recorded as 'other' for these two subjects. Many dressings detached when volunteers were away from the clinic and prior to returning for the assessments.
Measure: Number; unit: participants
Groups:
- AQUACEL® Foam Adhesive Dressing - Original Adhesive: Original adhesive
  AQUACEL® foam adhesive dressing
- AQUACEL® Foam Adhesive Dressing - Test Adhesive: Test adhesive
  AQUACEL® foam adhesive dressing
Arm/Group | AQUACEL® Foam Adhesive Dressing - Original Adhesive | AQUACEL® Foam Adhesive Dressing - Test Adhesive
Number analyzed (Participants) | 20 | 20
participants
  Arm Adhesion Excellent | 6 | 5
  Arm Adhesion Good | 1 | 0
  Arm Adhesion Average | 1 | 1
  Arm Adhesion Poor | 0 | 0
  Arm Adhesion Very Poor | 12 | 14
  Arm Dressing conformability Missing | 12 | 14
  Arm Dressing conformability Excellent | 6 | 5
  Arm Dressing conformability Good | 2 | 1
  Arm Ease of removal Missing | 12 | 14
  Arm Ease of removal very easy | 8 | 6
  Arm Comfort during removal Missing | 12 | 14
  Arm Comfort during removal Excellent | 6 | 6
  Arm Comfort during removal Good | 2 | 0
  Arm Dressing integrity missing | 12 | 14
  Arm Dressing integrity Excellent | 8 | 6
  Arm Adhesive residue on removal missing | 12 | 14
  Arm Adhesive residue on removal None | 6 | 6
  Arm Adhesive residue on removal Minimal | 2 | 0
  Back Adhesion Excellent | 0 | 1
  Back Adhesion Good | 2 | 1
  Back Adhesion Average | 2 | 0
  Back Dressing Conformability Excellent | 0 | 1
  Back Dressing Conformability Good | 2 | 1
  Back Dressing Conformability Average | 2 | 0
  Back Ease of Removal Very Easy | 4 | 2
  Back Comfort During Removal Excellent | 4 | 2
  Back Dressing Integrity Excellent | 4 | 2
  Back Adhesive Residue on Removal None | 4 | 2

2. Secondary Outcome: Safety - the Nature and Frequency of Adverse Events
Description: Safety will be determined by the nature and frequency of Adverse Events. Condition of the skin under and around the dressings along with the incidence of skin irritation will be assessed. The incidence and nature of all adverse events will be recorded.
  Condition of the skin was evaluated by the Skin Irritation Scale. The possible responses are doubtful reaction, weak positive reaction, strong positive reaction, extreme positive reaction, irritant reaction, and negative reaction.
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | AQUACEL® Foam Adhesive Dressing - Original Adhesive | AQUACEL® Foam Adhesive Dressing - Test Adhesive
Number analyzed (Participants) | 20 | 20
participants | 8 | 5

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | AQUACEL® Foam Adhesive Dressing - Original Adhesive | AQUACEL® Foam Adhesive Dressing - Test Adhesive
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AQUACEL® Foam Adhesive Dressing - Original Adhesive (N=20) | AQUACEL® Foam Adhesive Dressing - Test Adhesive (N=20)
Arm: General disorders and administration site conditions (Skin and subcutaneous tissue disorders) | 6 | 5
Arm: Application site pruritus (Skin and subcutaneous tissue disorders) | 6 | 5
Arm: Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 | 2
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1
Arm: Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1
Arm: Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Back:General disorders and administration site conditions (Skin and subcutaneous tissue disorders) | 2 | 3
Back: Application site pruritus (Skin and subcutaneous tissue disorders) | 2 | 3

LIMITATIONS AND CAVEATS:
Many dressings detached from the skin when the volunteers were at home/away from the clinic and prior to returning for the assessments. It was therefore not possible for the Investigator to give a rating for several parameters on several volunteers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality Agreement